CLINICAL TRIAL: NCT00323882
Title: A Phase I/II, Open-label, Dose-escalation Study of MDX-010 Administered Every 3 Weeks for 4 Doses in Patients With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: Study of MDX-010 in Patients With Metastatic Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-017 ST; CA184-017 (Other: BMS)
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Prostate Cancer; Neoplasm Metastasis
Keywords: Prostate Cancer; Oncology; Prostate; Cancer; Metastatic; Hormone; PSA; Metastatic Hormone-Refractory Prostate Cancer (HRPC)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDX-010 (Experimental)
  Interventions: Drug: MDX-010

INTERVENTIONS:
Drug: MDX-010 — selected dose administered IV every 3 weeks

SUMMARY:
Multicenter study in which patients with metastatic hormone refractory prostate cancer (HRPC), who have not had previous chemotherapy or immunotherapy treatments, received MDX-010 every 3 weeks for 4 doses (12 weeks total duration of induction). MDX-010 was administered at escalating dosage levels of 3, 5, and 10 mg/kg/dose infusions. At least 6 patients were to be enrolled in each dosage level. Patients who tolerated and responded to treatment or who had stable disease for 3 months or longer and who subsequently progressed during the follow up phase of the study had the option to receive additional treatment with MDX-010, up to 4 cycles. Patients were followed in the study for response up to 2 years and were followed for survival status for up to 5 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate
* Metastatic prostate cancer (positive bone scan or measurable disease)
* Total testosterone of less than 50 ng/dL, except for patients with prior orchiectomy, where testosterone does not need to be measured.
* Patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of antiandrogen and completion of a washout period and then observe disease progression.
* Patients must stop using any herbal product known to decrease PSA levels (eg., saw palmetto and PC-SPES) or any systemic or topical corticosteroid at least 4 weeks prior to screening. Progressive disease must be documented after discontinuation of these products.
* Progressive disease after androgen deprivation (or hormone therapy). For patients with measurable disease, progression will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. For patients with progression in, or without any measurable disease, a positive bone scan and elevated PSA will be required.
* Patients receiving bisphosphate therapy must have been on stable doses for at least 4 weeks with stable symptoms prior to enrollment.
* No prior chemotherapy or immunotherapy (tumor vaccine, cytokine, or growth factor given to control prostate cancer).
* Prior radiation therapy completed at least 4 weeks prior to enrollment. No prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.

Exclusion Criteria:

* Bone pain due to metastatic bone disease severe enough to require routine narcotic analgesic use.
* History of severe hypersensitivity reactions to drugs formulated with polysorbate 80.
* Patients with active autoimmune disease or a history of autoimmune disease that required systemic steroids or immunosuppressive medications, except for patients with vitiligo.
* Prior therapy with any anti-cytotoxic T-lymphocyte antigen 4 (anti-CTLA-4) antibody.
* Active infection requiring therapy.
* Concurrent medical condition requiring the use of systemic or topical corticosteroids; systemic or topical corticosteroids must be discontinued at least 4 weeks prior to enrollment. The use of inhaled corticosteroids is acceptable.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (13):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Josephine Ford Cancer Center-Downriver, Brownstown, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center-West Bloomfield, West Bloomfield, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Sun BL. Immunotherapy in treatment of metastatic prostate cancer: An approach to circumvent immunosuppressive tumor microenvironment. Prostate. 2021 Nov;81(15):1125-1134. doi: 10.1002/pros.24213. Epub 2021 Aug 26. PMID 34435699
- [Derived] Iwama S, De Remigis A, Callahan MK, Slovin SF, Wolchok JD, Caturegli P. Pituitary expression of CTLA-4 mediates hypophysitis secondary to administration of CTLA-4 blocking antibody. Sci Transl Med. 2014 Apr 2;6(230):230ra45. doi: 10.1126/scitranslmed.3008002. PMID 24695685
- [Derived] Slovin SF, Higano CS, Hamid O, Tejwani S, Harzstark A, Alumkal JJ, Scher HI, Chin K, Gagnier P, McHenry MB, Beer TM. Ipilimumab alone or in combination with radiotherapy in metastatic castration-resistant prostate cancer: results from an open-label, multicenter phase I/II study. Ann Oncol. 2013 Jul;24(7):1813-1821. doi: 10.1093/annonc/mdt107. Epub 2013 Mar 27. PMID 23535954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated January 2006; Primary endpoint last visit September 2009; follow up period last visit July 2013 with data cut off September 2013. Male patients with castrate-resistant prostate cancer (CRPC) who met study criteria were enrolled.
Pre-assignment Details: 75 participants enrolled and were assigned to treatment; 71 were treated. Reasons for the 4 participants not receiving treatment were not specified by the investigators. Ipilimumab was administered at escalating dosage levels of 3, 5, and 10 mg/kg/dose.
Groups:
- Ipilimumab Monotherapy 3 mg/kg: A single dose of 3 mg/kg ipilimumab was administered over 90 minutes intravenously (IV) on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. Those participants with a clinical response of stable disease (SD) or conflicting disease response assessment (CDRA) at the end of the induction period could have received additional treatment up to a total of 16 doses in the maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Ipilimumab Monotherapy 5 mg/kg: A single dose of 5 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses (induction). Those participants with a clinical response of SD or CDRA at the end of induction could have received additional treatment up to a total of 16 doses (maintenance). The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Ipilimumab Monotherapy 10 mg/kg: A single dose of 10 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. Those participants with a clinical response of SD or CDRA at the end of induction could have received additional treatment up to a total of 16 doses in the maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Ipilimumab 3 mg/kg + XRT Combination Therapy: A single dose of 3 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. In addition, participants received a single dose of 800 rads (8 Gray) of focal radiotherapy (XRT) to each target lesion within 48 hours before the first infusion of ipilimumab during the induction period. According to Response Evaluation Criteria in Solid Tumors (RECIST), target or measurable lesions were defined as lesions that could be accurately measured in at least one dimension (longest diameter recorded) as ≥ 10 mm with spiral computed tomography (CT). Those participants with a clinical response of SD or CDRA at the end of induction could have received additional treatment up to a total 16 doses in the maintenance period. Radiotherapy was not administered during maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Ipilimumab 10 mg/kg + XRT Combination: A single dose of 10 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. In addition, participants received a single dose of 800 rads (8 Gray) of focal XRT to each target lesion within 48 hours before the first infusion of ipilimumab in the induction period. According to RECIST, target or measurable lesions were defined as lesions that could be accurately measured in at least one dimension (longest diameter recorded) as ≥ 10 mm with spiral CT. Those participants with a clinical response of SD or CDRA at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. Radiotherapy was not administered during maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
Period: Overall Study
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Started | 8 | 6 | 16 | 7 | 34
Completed | 0 | 0 | 3 | 0 | 2
Not Completed | 8 | 6 | 13 | 7 | 32
Not completed — Adverse Event | 2 | 1 | 1 | 1 | 3
Not completed — Disease Progression | 6 | 4 | 10 | 5 | 22
Not completed — Death | 0 | 1 | 1 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study therapy.
Groups:
- Ipilimumab Monotherapy 3 mg/kg: A single dose of 3 mg/kg ipilimumab was administered over 90 minutes intravenously (IV) on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. Those participants with a clinical response of stable disease (SD) or conflicting disease response assessment (CDRA) at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Ipilimumab Monotherapy 5 mg/kg: A single dose of 5 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses (induction). Those participants with a clinical response of SD or CDRA at the end of induction could have received additional treatment up to a total of 16 doses in the maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Ipilimumab 3 mg/kg + XRT Combination Therapy: A single dose of 3 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. In addition, participants received a single dose of 800 rads (8 Gray) of focal radiotherapy (XRT) to each target lesion within 48 hours before the first infusion of ipilimumab during the induction period. According to RECIST, target or measurable lesions were defined as lesions that could be accurately measured in at least one dimension (longest diameter recorded) as ≥ 10 mm with spiral computed tomography (CT). Those participants with a clinical response of SD or CDRA at the end of induction could have received additional treatment up to a total 16 doses in the maintenance period. Radiotherapy was not administered during maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination | Total
Number analyzed (Participants) | 8 | 6 | 16 | 7 | 34 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.1) | 58.2 (5.6) | 65.2 (7.7) | 67.6 (8.5) | 65.7 (9.1) | 65.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 16 | 7 | 34 | 71
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Black | 0 | 0 | 0 | 1 | 3 | 4
  White | 8 | 6 | 16 | 6 | 30 | 66
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 16 | 7 | 34 | 71
Mean Prostate-Specific Antigen (PSA) in ng/mL [Mean (Standard Deviation); unit: ng/mL] — PSA is measured in nanograms per milliliter (ng/mL).
  ng/mL | 121.6 (140.2) | 48.8 (43.9) | 302.7 (521.2) | 66.6 (68.1) | 250.1 (324.1) | 212.9 (346.5)
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants] — ECOG performance: 0= Fully active, able to carry on all pre-disease performance without restriction;1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or Chair; 5=Dead
  participants
    ECOG PS 0 | 5 | 5 | 10 | 4 | 9 | 33
    ECOG PS 1 | 3 | 1 | 6 | 2 | 22 | 34
    ECOG PS 2 | 0 | 0 | 0 | 1 | 0 | 1
    ECOG PS Not Reported | 0 | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious AEs (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Immune-related AEs - Treated Participants
Description: AEs graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling, Gr 5=Death. Related=relationship to study drug reported as certain, probable, possible, or missing. Immune-related AE (irAE) was defined as a clinically significant AE of any organ that is associated with drug exposure, of unknown etiology, and is consistent with an immune-mediated mechanism. Day 1=first day of study treatment.
Time Frame: Day 1 to last day of study treatment (+70 days) up to 2 years
Population: All participants in the study who received either ipilimumab or radiation were analyzed.
Measure: Number; unit: participants
Groups:
- Ipilimumab Monotherapy 3 mg/kg: A single dose of 3 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. Those participants with a clinical response of SD or CDRA at the end induction period could have received additional treatment up to a total of 16 doses in the maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 8 | 6 | 16 | 7 | 34
participants
  SAE | 3 | 2 | 9 | 2 | 19
  Drug-Related SAE | 2 | 1 | 7 | 2 | 7
  AEs leading to discontinuation | 2 | 2 | 7 | 3 | 13
  Related-AEs leading to discontinuation | 2 | 2 | 6 | 3 | 8
  Grade 3-4 AE | 2 | 5 | 12 | 3 | 20
  Related AE (Any Grade) | 8 | 5 | 16 | 6 | 29
  Grade 3-4 Related AE | 2 | 3 | 10 | 3 | 13
  irAE (Any Grade) | 6 | 5 | 16 | 4 | 24
  Grade 3-4 irAE | 1 | 3 | 10 | 3 | 6

2. Secondary Outcome: Number of Participants With Best Overall PSA Response by Category - PSA Evaluable Participants
Description: Best Overall PSA response per investigator, using NCI PSA Working Group: PSA with CR or PR at any time after treatment initiation and was confirmed at least 4 weeks after the first measurement. PSA reference=PSA measured immediately prior to treatment. CR=PSA concentration < 2 nanograms per milliliter (ng/mL), confirmed at least 4 weeks after 1st value; PR=PSA concentration ≤ 50% of PSA reference, confirmed at least 4 weeks after 1st value; Unconfirmed=not confirmed by repeat measurements; SD=No change from PSA reference value; PD = If PSA nadir was ≥ 100% of the reference value: PSA ≥ 125% of PSA reference and with a difference of absolute value of ≥ 5 ng/mL; If PSA nadir was < 100% and ≥ 50% of the reference value: PSA ≥ 125% of PSA nadir and with a difference of absolute value of ≥ 5 ng/mL: If PSA nadir was < 50% of the reference value: PSA ≥ 150% of PSA nadir and with a difference of absolute value of ≥ 5 ng/mL.
Time Frame: Day 1 to last day of study treatment (+70 days) up to 2 years
Population: PSA-evaluable participants, including all participants in cohorts with monotherapy and with radiotherapy who received any ipilimumab and had a baseline PSA, were analyzed.
Measure: Number; unit: participants
Groups:
- Ipilimumab Monotherapy 3 mg/kg: A single dose of 3 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. Those participants with a clinical response of SD or CDRA at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 8 | 6 | 16 | 6 | 34
participants
  Complete Response (CR) | 0 | 0 | 1 | 0 | 2
  Partial Response (PR) | 2 | 1 | 3 | 2 | 2
  Unconfirmed Partial Response | 0 | 0 | 2 | 0 | 2
  Stable Disease (SD) | 3 | 4 | 6 | 2 | 14
  Progressive Disease (PD) | 3 | 1 | 3 | 2 | 11
  Unknown | 0 | 0 | 1 | 0 | 3

3. Secondary Outcome: Number of Participants With Best Overall Tumor Response by Category - Tumor Evaluable Participants
Description: For those with measurable disease, tumor response based upon tumor lesions (per investigator) using Response Evaluation Criteria in Solid Tumors (RECIST). Best Overall=Participants with a best tumor response of CR or PR at anytime during the study. CR=Disappearance of all target lesions; PR=At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference, baseline sum LD. For a status of CR or PR, changes in tumor measurements were confirmed by repeat studies no less than 4 weeks after the criteria for response were first met; Unconfirmed=not confirmed by repeat measurements; SD=Neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum LD since the treatment started; PD=At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Day 1 to last day of study treatment (+70 days) up to 2 years
Population: Tumor-evaluable participants, including all participants in cohorts with monotherapy and with radiotherapy who received any ipilimumab and had measurable disease at baseline, were analyzed.
Measure: Number; unit: participants
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 1 | 1 | 8 | 2 | 20
participants
  Complete Response | 0 | 0 | 1 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0
  Unconfirmed Partial Response | 0 | 0 | 1 | 0 | 1
  Stable Disease | 1 | 1 | 1 | 1 | 5
  Progressive Disease | 0 | 0 | 3 | 1 | 5
  Unknown | 0 | 0 | 2 | 0 | 9

4. Secondary Outcome: Time to PSA Response at Day 85 in Participants With Complete Response (CR) or Confirmed Partial Response (PR) at Day 85
Description: Time to PSA response was measured in months. Time to PSA response was analyzed in those participants with CR or PR at Day 85. CR=PSA concentration < 2 ng/mL, confirmed at least 4 weeks after 1st value; PR=PSA concentration ≤ 50% of PSA reference, confirmed at least 4 weeks after 1st value.
Time Frame: Day 1 to Day 85
Population: All participants in cohorts with monotherapy and with radiotherapy who received any ipilimumab, had a baseline PSA, and had a confirmed Complete Response (CR) or Partial Response (PR) at Day 85.
Measure: Median (Full Range); unit: Months
Groups:
- Ipilimumab 10 mg/kg + XRT Combination (Prior Chemotherapy); Ipilimumab 10 mg/kg + XRT Combination (Chemotherapy Naive): A single dose of 10 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. In addition, participants received a single dose of 800 rads (8 Gray) of focal XRT to each target lesion within 48 hours before the first infusion of ipilimumab in the induction period. According to RECIST, target or measurable lesions were defined as lesions that could be accurately measured in at least one dimension (longest diameter recorded) as ≥ 10 mm with spiral CT. Those participants with a clinical response of SD or CDRA at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. Radiotherapy was not administered during maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination (Prior Chemotherapy) | Ipilimumab 10 mg/kg + XRT Combination (Chemotherapy Naive)
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 2 | 2
Months | 1.41 [1.41 to 1.41] | 1.54 [1.54 to 1.54] | 1.4 [0.9 to 2.3] |  | 1.1 [0.8 to 1.5] | 1.1 [0.8 to 1.4]

5. Secondary Outcome: Overall Tumor Response Rate in 10 mg/kg Ipilimumab Monotherapy and Ipilimumab/XRT Combination Therapy
Description: Tumor response rate was defined as the number of participants with a best response of partial or complete response divided by the total number of tumor evaluable participants. Overall Tumor Response was defined as participants with a tumor response of CR or PR at anytime during the study. CR=Disappearance of all target lesions; PR=At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference, baseline sum LD. For a status of CR or PR, changes in tumor measurements were confirmed by repeat studies no less than 4 weeks after the criteria for response were first met
Time Frame: Day 1 to last day of study treatment (+70 days) up to 2 years
Population: All participants in cohorts with 10 mg/kg ipilimumab monotherapy and with 10 mg/kg ipilimumab combination therapy with XRT who received any ipilimumab and had a baseline PSA, were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ipilimumab 10 mg/kg + XRT Combination (Prior Chemotherapy): In those who received chemotherapy prior to enrolling in this study, a single dose of 10 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. In addition, participants received a single dose of 800 rads (8 Gray) of focal XRT to each target lesion within 48 hours before the first infusion of ipilimumab in the induction period. According to RECIST, target or measurable lesions were defined as lesions that could be accurately measured in at least one dimension (longest diameter recorded) as ≥ 10 mm with spiral CT. Those participants with a clinical response of SD or CDRA at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. Radiotherapy was not administered during maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
- Ipilimumab 10 mg/kg + XRT Combination (Chemotherapy Naive): In those participants who had received no chemotherapy prior to the study, a single dose of 10 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. In addition, participants received a single dose of 800 rads (8 Gray) of focal XRT to each target lesion within 48 hours before the first infusion of ipilimumab in the induction period. According to RECIST, target or measurable lesions were defined as lesions that could be accurately measured in at least one dimension (longest diameter recorded) as ≥ 10 mm with spiral CT. Those participants with a clinical response of SD or CDRA at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. Radiotherapy was not administered during maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
Arm/Group | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 10 mg/kg + XRT Combination (Prior Chemotherapy) | Ipilimumab 10 mg/kg + XRT Combination (Chemotherapy Naive)
Number analyzed (Participants) | 8 | 16 | 4
percentage of participants | 12.5 [0.3 to 52.7] | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: PSA Response Rate at Day 85 and Overall PSA Response Rate in 10 mg/kg Monotherapy and Combination Therapy
Description: PSA response rate was defined as the number of participants with a PSA response (PR or CR) divided by the total number of PSA evaluable participants. PSA response at Day 85, as reported by the investigator, was defined as a PSA concentration < 50% of the PSA reference value occurring on or before Day 85 and this response was confirmed at least 4 weeks after the first determination. The PSA reference value was the PSA concentration measured immediately prior to treatment. Overall Response is < 50% of the PSA reference value occurring anytime after treatment was initiated and this response was confirmed at least 4 weeks after the first determination. Complete response=PSA concentration < 2 ng/mL, confirmed at least 4 weeks after first value; Partial response=PSA concentration ≤ 50% of PSA reference value, confirmed at least 4 weeks after first determination.
Time Frame: Day 85, Day 1 to last day of study treatment (+70 days) up to 2 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ipilimumab 10 mg/kg + XRT Combination (Chemotherapy Naive): In those participants with no prior chemotherapy, a single dose of 10 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses in the induction period. In addition, participants received a single dose of 800 rads (8 Gray) of focal XRT to each target lesion within 48 hours before the first infusion of ipilimumab in the induction period. According to RECIST, target or measurable lesions were defined as lesions that could be accurately measured in at least one dimension (longest diameter recorded) as ≥ 10 mm with spiral CT. Those participants with a clinical response of SD or CDRA at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. Radiotherapy was not administered during maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
Arm/Group | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 10 mg/kg + XRT Combination (Prior Chemotherapy) | Ipilimumab 10 mg/kg + XRT Combination (Chemotherapy Naive)
Number analyzed (Participants) | 16 | 21 | 13
percentage of participants
  PSA Response Rate at Day 85 | 18.8 [4.0 to 45.6] | 9.5 [1.2 to 30.4] | 15.4 [1.9 to 45.4]
  Overall PSA Response Rate | 25.0 [7.3 to 52.4] | 9.5 [1.2 to 30.4] | 15.4 [1.9 to 45.4]

7. Primary Outcome: Number of Participants With Best PSA Response at Day 85 by Category - PSA Evaluable Participants
Description: Response by investigator using National Cancer Institute (NCI) PSA Working Group recommendations= PSA < 50% of PSA reference value occurring on or before Day 85; response confirmed at least 4 weeks after the first measurement. PSA reference=PSA measured immediately prior to treatment. Complete response (CR)=PSA < 2 nanograms per milliliter (ng/mL), confirmed at least 4 weeks after 1st value; Partial response (PR)=PSA ≤ 50% of PSA reference, confirmed at least 4 weeks after 1st value; Unconfirmed=not confirmed by repeat measurements; Stable disease(SD)=No change from PSA reference; Progressive disease (PD) defined: If PSA nadir was ≥ 100% of the reference: PSA ≥ 125% of PSA reference and with a difference of absolute value of ≥ 5 ng/mL; If PSA nadir was < 100% and ≥ 50% of the reference: PSA ≥ 125% of PSA nadir and with a difference of absolute value of ≥ 5 ng/mL: If PSA nadir was < 50% of the reference: PSA ≥ 150% of PSA nadir and with a difference of absolute value of ≥ 5 ng/mL.
Time Frame: Day 85
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 8 | 6 | 16 | 6 | 34
participants
  Complete Response | 0 | 0 | 1 | 0 | 1
  Partial Response | 1 | 1 | 2 | 0 | 3
  Unconfirmed Partial Response | 0 | 0 | 2 | 0 | 1
  Stable Disease | 4 | 4 | 7 | 4 | 14
  Progressive Disease | 3 | 1 | 3 | 2 | 11
  Unknown | 0 | 0 | 1 | 0 | 4

8. Secondary Outcome: Number of Participants Who Died by Date of Primary Analysis and by Date of Completion of Follow Up - All Treated Participants
Description: Primary analysis was conducted on data from Day 1 up to 2 years post treatment, data available as of September 2009. Final Follow-Up analysis was conducted on data up to 5 years post treatment, data available as of September 2013 (minimum time of eligibility 54 months to a maximum of 85 months). Primary causes of deaths are listed under each timepoint.
Time Frame: Day 1 to 5 years post treatment
Population: Treated participants population included all participants in the study who received either ipilimumab or radiation.
Measure: Number; unit: participants
Groups:
- All Treated Participants: All participants in all treatment arms combined.
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination | All Treated Participants
Number analyzed (Participants) | 8 | 6 | 16 | 7 | 34 | 71
participants
  Total Deaths at Primary Analysis | 5 | 4 | 7 | 3 | 18 | 37
  Maliginant Disease | 0 | 0 | 0 | 0 | 3 | 3
  Prostate Cancer | 1 | 3 | 4 | 3 | 10 | 21
  Toxicity | 0 | 1 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 2 | 2
  Unknown | 3 | 0 | 3 | 0 | 3 | 9
  No cause specified | 1 | 0 | 0 | 0 | 0 | 1
  Total Deaths at Completion of Follow Up | 7 | 6 | 11 | 7 | 29 | 60
  Malignant Disease | 0 | 0 | 0 | 0 | 3 | 3
  Prostate Cancer | 1 | 4 | 6 | 4 | 13 | 28
  Toxicity | 0 | 1 | 0 | 0 | 0 | 1
  Other | 0 | 1 | 1 | 0 | 5 | 7
  Unknown | 5 | 0 | 4 | 3 | 8 | 20
  No cause specified | 1 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Overall Survival at Completion of Follow Up Period - Treated Participants
Description: Overall Survival (OS) was defined as the time from the first date of study treatment until the date of death and was measured in months. For those participants who have not died, OS was censored at the last date the participant was known to be alive. Completion of follow-up for OS was a minimum time of eligibility 54 months to a maximum of 85 months.
Time Frame: Day 1 to 5 years post treatment
Population: All participants in cohorts with monotherapy and with radiotherapy who received any ipilimumab were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Treated Participants: All treatment groups are combined to show total overall survival at completion of Follow Up.
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination | All Treated Participants
Number analyzed (Participants) | 8 | 6 | 16 | 7 | 34 | 71
Months | 22.5 [11.5 to 59.9] | 36.3 [28.0 to 41.8] | 26.6 [8.6 to 49.9] | 18.2 [10.0 to 24.7] | 9.7 [5.6 to 16.4] | 17.4 [11.5 to 24.7]

10. Secondary Outcome: Number of Participants With On-Study Hematology Laboratory Tests Worst Common Terminology Criteria (CTC) Grade - Treated Participants
Description: NCI CTC version(v) 3.0 was used to determine Grade (Gr). Screening was Day -28 to Day -1. On-study laboratories were reported after the first dose date, every 21 days during a treatment cycle, and within 70 days of last dose of study therapy (ie, Days 1, 22, 43, 64, 85, etc). Hemoglobin grams per liter (g/L): Gr 1: 10.0 - less than (<) lower limit of normal (LLN); Gr 2: 8.0 - < 10.0; Gr 3: 6.5 - < 8.0; Gr 4: < 6.5. White blood cells(WBC) 10^9 cells per liter (c/L): Gr1: 3.0 - < LLN; Gr 2: 2.0 - < 3.0; Gr 3: 1.0 - < 2.0; Gr4: < 1.0. Lymphocytes (absolute) 10^9 c/L: Gr1: 0.8 - < 1.5; Gr 2: 0.5 - < 0.8; Gr 3): 0.2 - < 0.5; Gr 4: < 0.2. Neutrophils (absolute) 10^9 c/L: Gr 1: 1.5 - < 2.0; Gr 2: 1.0 - < 1.5; Gr 3: 0.5 - < 1.0; Gr 4: < 0.5. Platelets 10^9 c/L: Gr 1: 75.0 - < lower limits of normal (LLN); Gr 2: 50.0 - < 75.0; Gr 3: 25.0 - < 50.0; Gr 4: < 25.0.
Time Frame: Day 1 to last day of study treatment (+70 days) up to 2 years
Population: All participants in the study who received either ipilimumab or radiation and had a laboratory measurement were analyzed.
Measure: Number; unit: participants
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 8 | 5 | 15 | 6 | 34
participants
  WBC Grade 1-4 (n=8, 5, 15, 6, 34) | 0 | 0 | 0 | 1 | 2
  WBC Grade 3-4 (n=8, 5, 15, 6, 34) | 0 | 0 | 0 | 0 | 0
  Neutrophils Grade 1-4 (n=8, 5, 15, 6, 34) | 2 | 0 | 0 | 1 | 2
  Neutrophils Grade 3-4 (n=8, 5, 15, 6, 34) | 0 | 0 | 0 | 0 | 0
  Platelets Grade 1-4 (n=8, 5, 15, 6, 34) | 0 | 0 | 1 | 1 | 2
  Platelets Grade 3-4 (n=8, 5, 15, 6, 34) | 0 | 0 | 0 | 0 | 0
  Hemoglobin Grade 1-4 (n=8, 5, 15, 6, 34) | 7 | 4 | 12 | 6 | 28
  Hemoglobin Grade 3-4 (n=8, 5, 15, 6, 34) | 0 | 0 | 1 | 0 | 6
  Lymphocytes Grade 1-4 (n=8, 5, 15, 6, 34) | 7 | 3 | 12 | 5 | 31
  Lymphocytes Grade 3-4 (n=8, 5, 15, 6, 34) | 0 | 0 | 2 | 1 | 3

11. Secondary Outcome: Number of Participants With On-Study Serum Chemistry Laboratory Tests Worst Common Terminology Criteria (CTC) Grade - Treated Participants
Description: CTC v3.0 used. On-study serum chemistry laboratories were reported after first dose date, every 21 days during a treatment cycle, and within 70 days of last dose of study therapy (ie, Days 1, 22, 43, 64, 85, etc). Alanine Aminotransferase (ALT) Units per Liter (U/L) Gr 1: > 1.0 - 2.5 * upper limits of normal (ULN); Gr 2: > 2.5 - 5.0 * ULN; Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Aspartate Aminotransferase (AST) U/L: Gr 1: > 1.0 - 2.5 * ULN; Gr 2: > 2.5 - 5.0 * ULN; Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Total Bilirubin micromoles per liter (µmol/L): Gr 1: > 1.0 - 1.5 * ULN; Gr 2: > 1.5 - 3.0 * ULN; Gr 3: > 3.0 - 10.0 * ULN; Gr 4: > 10.0 * ULN. Alkaline Phosphatase U/L: Gr 1: > 1.0 - 2.5 * ULN; Gr 2: > 2.5 - 5.0 * ULN; Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Amylase U/L: Gr1: > 1.0 - 1.5 * ULN; Gr 2: > 1.5 - 2.0 * ULN; Gr 3: > 2.0 - 5.0 * ULN; Gr4: > 5.0 * ULN. Creatinine µmol/L: Gr1: > 1.0 - 1.5*ULN; Gr2: > 1.5 - 3.0*ULN; Gr3: > 3.0 - 6.0*ULN; Gr4: > 6.0*ULN.
Time Frame: Day 1 to last day of study treatment (+70 days) up to 2 years
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 8 | 5 | 15 | 6 | 34
participants
  ALT Grade 1-4 (n=8,5,15,6,34) | 0 | 2 | 7 | 2 | 10
  ALT Grade 3-4 (n=8,5,15,6,34) | 0 | 1 | 2 | 0 | 1
  AST Grade 1-4 (n=8,5,15,6,34) | 0 | 2 | 6 | 2 | 8
  AST Grade 3-4 (n=8,5,15,6,34) | 0 | 1 | 2 | 0 | 0
  Bilirubin Grade 1-4 (n=8,5,15,6,34) | 0 | 0 | 2 | 1 | 1
  Bilirubin Grade 3-4 (n=8,5,15,6,34) | 0 | 0 | 0 | 0 | 0
  Phosphatase Grade 1-4 (n=8,5,15,6,34) | 3 | 4 | 7 | 5 | 21
  Phosphatase Grade 3-4 (n=8,5,15,6,34) | 0 | 0 | 1 | 1 | 5
  Amylase Grade 1-4 (n=8,5,15,6,34) | 2 | 3 | 4 | 0 | 4
  Amylase Grade 3-4 (n=8,5,15,6,34) | 0 | 0 | 0 | 0 | 1
  Creatinine Grade 1-4 (n=8,5,15,6,34) | 0 | 0 | 4 | 1 | 5
  Creatinine Grade 3-4 (n=8,5,15,6,34) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities at Baseline and During Treatment Period - Treated Participants
Description: 12 Lead Electrocardiograms (ECGs) were performed at screening (Day -28 to Day -1), and on Day 85 during a treatment cycle, and at the end of treatment period. Clinically significant abnormalities could include atrial fibrillation, anterior fascicular block, marked sinus bradycardia, possible lateral infarct, and T-wave abnormality (other potential abnormalities were not excluded from consideration).
Time Frame: Baseline up to 2 years
Population: All participants in the study who received either ipilimumab or radiation and had an ECG were analyzed.
Measure: Number; unit: participants
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 8 | 6 | 15 | 7 | 31
participants
  ECG Abnormalities at Baseline (n=8, 6, 15, 7, 31) | 0 | 0 | 2 | 0 | 0
  ECG Abnormalities During Treatment (n=4,3,11,4,20) | 0 | 0 | 2 | 0 | 0

13. Secondary Outcome: Number of Participants Positive for Human Anti-Human Antibodies (HAHA) - Treated Participants
Description: HAHA was measured by electrochemiluminescent (ECL) immunoassay for the detection of antibodies in human heparin plasma. Testing was performed on Days 1 (prior to ipilimumab infusion), 64, 85, and at completion of treatment.
Time Frame: Day 1 up to 2 years
Population: All participants in the study who received either ipilimumab or radiation and had a measurement were analyzed.
Measure: Number; unit: participants
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Number analyzed (Participants) | 8 | 6 | 16 | 7 | 34
participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to last day of study treatment (+70 days) up to 2 years
Groups:
- Ipilimumab Monotherapy 5 mg/kg: A single dose of 5 mg/kg ipilimumab was administered over 90 minutes IV on Days 1, 22, 43, and 64 for a total of 4 doses (induction). Those participants with a clinical response of SD or CDRA at the end of induction period could have received additional treatment up to a total of 16 doses in the maintenance period. The length of time on study for an individual could be up to 2 years. Follow up for survival status was for up to 5 years after enrollment.
Arm/Group | Ipilimumab Monotherapy 3 mg/kg | Ipilimumab Monotherapy 5 mg/kg | Ipilimumab Monotherapy 10 mg/kg | Ipilimumab 3 mg/kg + XRT Combination Therapy | Ipilimumab 10 mg/kg + XRT Combination
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/6 | 9/16 | 2/7 | 19/34
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 16/16 | 6/7 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab Monotherapy 3 mg/kg (N=8) | Ipilimumab Monotherapy 5 mg/kg (N=6) | Ipilimumab Monotherapy 10 mg/kg (N=16) | Ipilimumab 3 mg/kg + XRT Combination Therapy (N=7) | Ipilimumab 10 mg/kg + XRT Combination (N=34)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Hypophysitis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 4 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 4
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab Monotherapy 3 mg/kg (N=8) | Ipilimumab Monotherapy 5 mg/kg (N=6) | Ipilimumab Monotherapy 10 mg/kg (N=16) | Ipilimumab 3 mg/kg + XRT Combination Therapy (N=7) | Ipilimumab 10 mg/kg + XRT Combination (N=34)
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 3
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 5
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 6 | 3 | 13
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 3 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 2
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 2 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 1 | 6
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 2 | 1 | 2
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 6 | 3 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 10 | 1 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 5 | 4 | 10
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 6 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Dysphoria (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 5 | 9 | 4 | 19
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lipase (Investigations) | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 3 | 1 | 7
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 2 | 1 | 2
Nocturia (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 2 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2 | 8
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 2
Blood amylase increased (Investigations) | 0 | 2 | 0 | 0 | 2
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 2 | 0 | 5
Pyrexia (General disorders) | 1 | 2 | 2 | 1 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 7 | 5 | 7
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 13 | 3 | 17
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1
Infusion related reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 1 | 0 | 2
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 2 | 0 | 0
Euthyroid sick syndrome (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mucosal exfoliation (General disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 1 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0 | 6
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 8 | 4 | 15
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 6 | 0 | 4
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid factor increased (Investigations) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the small number of participants who underwent more than 4 doses of treatment (induction period) and the exploratory nature of this study, not all of the secondary objectives were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.